CLINICAL TRIAL: NCT03836040
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Erenumab in Children (6 to < 12 Years) and Adolescents (12 to < 18 Years) With Episodic Migraine (OASIS PEDIATRIC [EM])
Brief Title: Efficacy and Safety of Erenumab in Pediatric Participants With Episodic Migraine
Acronym: OASIS(EM)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150125; 2023-504930-23 (EudraCT Number)
Record Dates: First submitted 2019-01-29; First posted 2019-02-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Migraine
Keywords: Migraine; Headache; Prevention; Pediatric; Episodic Migraine
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose level 1 (Experimental): Participants will be randomized to one of two doses determined by their body weight at Day 1. Participants who enrolled under the original protocol or protocol amendment 1 will be identified as group 1. Those enrolled under protocol amendment 2 will be identified as group 2.
  Interventions: Drug: Erenumab Dose 1; Drug: Erenumab Dose 2
- Dose level 2 (Experimental): Participants will be randomized to one of two doses determined by their body weight at Day 1. Participants who enrolled under the original protocol or protocol amendment 1 will be identified as group 1. Those enrolled under protocol amendment 2 will be identified as group 2.
  Interventions: Drug: Erenumab Dose 2; Drug: Erenumab Dose 3
- Placebo (Placebo Comparator): Participants will be randomized to a placebo comparator.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Erenumab Dose 1 — Participants in the low body-weight group at day 1 and who are randomized to Dose Level 1 will receive this dose.
  Other Names: AMG334; Aimovig®
  Arms: Dose level 1
Drug: Erenumab Dose 2 — Participants in the low body-weight group at day 1 who are randomized to Dose Level 2 and subjects in the high body-weight group at day 1 who are randomized to Dose Level 1 will receive this dose.
  Other Names: AMG 334; Aimovig®
  Arms: Dose level 1; Dose level 2
Drug: Erenumab Dose 3 — Participants in the high body-weight group at day 1 who are randomized to Dose Level 2 will receive this dose.
  Other Names: AMG 334; Aimovig®
  Arms: Dose level 2
Other: Placebo — Placebo matching dose for erenumab dose 1, 2 and 3.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of erenumab in migraine prevention in children (6 to <12 years) and adolescents (12 to <18 years) with episodic migraine. The study hypothesis is that in pediatric participants with episodic migraine, the combined erenumab dose group has a greater reduction from baseline to week 9 through week 12 (month 3) in monthly migraine days (MMDs) when compared with placebo in the double-blind treatment phase (DBTP).

DETAILED DESCRIPTION:
This study is a Phase 3, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of erenumab in migraine prevention in children (6 to <12 years) and adolescents (12 to <18 years) with episodic migraine.

The trial consists of four phases: screening (up to 3 weeks of initial screening and a 4-week prospective baseline phase); the DBTP (24 weeks for Group 1 participants; 12-weeks for Group 2 participants) in which participants receive placebo or Erenumab dose 1, dose 2 or dose 3 (based on participant's body weight) via subcutaneous injection once a month; the optional dose level blinded extension phase (40 weeks), in which all participants are assigned to receive dose 1, dose 2 or dose 3 of Erenumab; and a 12 weeks safety follow-up phase (16 weeks after the last dose of investigational drug).

The study intends to enroll 436 participants (376 adolescents and up to 60 children).

ELIGIBILITY:
* Inclusion Criteria

  * Children (6 to less than 12 years of age) or adolescent (12 to less than 18 years of age) at the time of signing, if developmentally appropriate, the formal assent to participate to the study.
  * Participant's parent or legal representative has provided written informed consent before initiation of any study-specific activities/procedures.
  * History of migraine (with or without aura) for greater than or equal to 12 months before screening according to the IHS Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2013) based on medical records and/or participant self-report or parents' or legal representative's report.
  * The following ICHD-3 specifications for pediatric migraine (participants aged less than 18 years), should be considered for the diagnosis of migraine:
  * Attacks may last 2 to 72 hours.
  * Migraine headache is more often bilateral than in adults; unilateral pain usually emerges in late adolescence or early adult life.
  * Migraine headache is usually frontotemporal. Occipital headache in children is rare and calls for diagnostic caution.
  * A subset of otherwise typical participants have facial location of pain, which is called 'facial migraine' in the literature; there is no evidence that these participants form a separate subgroup of migraine participants.
  * In young children, photophobia and phonophobia may be inferred from their behavior.
  * History of less than 15 headache days per month of which greater than or equal to 4 headache days were assessed by the participant as migraine days in each of the 3 months prior to screening (refer to Section 5.6 for definition of migraine day).
* Criteria to be assessed prospectively during the 4-week baseline phase and confirmed before randomizing the participant into the DBTP:

  * Migraine frequency: greater than or equal 4 and less than 15 migraine days based on the eDiary data during the last 28 days of the baseline phase if greater than 28 days in duration
  * Headache frequency: less than 15 headache days based on the eDiary data during the last 28 days of the baseline phase if greater than 28 days in duration.
  * Demonstrated at least 80% compliance with the eDiary based on the last 28 days of the baseline period, if greater than 28 days in duration (eg, completing eDiary items for at least 23 out of the last 28 days of the baseline phase).
* Exclusion Criteria

  • History of cluster headache or hemiplegic migraine headache.
* No therapeutic response with greater than 2 of the following 10 medication categories for prophylactic treatment of migraine after an adequate therapeutic trial. These medication categories are:

  * Category 1: beta blockers (eg, propranolol, atenolol, bisoprolol, metoprolol, nadolol, nebivolol, pindolol, timolol)
  * Category 2: tricyclic antidepressants (eg, amitriptyline, nortriptyline, protriptyline)
  * Category 3: topiramate
  * Category 4: divalproex sodium, sodium valproate
  * Category 5: serotonin-norepinephrine reuptake inhibitors (eg, venlafaxine, desvenlafaxine, duloxetine, milnacipran)
  * Category 6: cyproheptadine
  * Category 7: flunarizine, cinnarizine
  * Category 8: botulinum toxin
  * Category 9: lisinopril/candesartan
  * Category 10: medications targeting the CGRP pathway.
* No therapeutic response is defined as no reduction in headache frequency, duration, or severity after administration of the medication for at least 6 weeks at the generally-accepted therapeutic dose(s) based on the investigator's assessment.
* The following scenarios do not constitute lack of therapeutic response:

  * Lack of sustained response to a medication.
  * Partial, suboptimal response to a medication.
  * Failure to tolerate a therapeutic dose.
  * Evidence of drug or alcohol abuse or dependence within 12 months before screening, based on medical records, participant self-report, or positive urine drug test performed during screening (with the exception of prescribed medications such as opioids or barbiturates).
  * Human immunodeficiency virus (HIV) infection by history.
  * History of seizure disorder or other significant neurological disorder other than migraine. Note: a single childhood febrile seizure is not exclusionary.
  * History of major psychiatric disorder (such as schizophrenia, schizoaffective disorder, bipolar disorder, obsessive-compulsive disorder, or pervasive developmental disorder), or current evidence of major depressive disorder based on a patient health questionnaire-9 modified for adolescents (PHQ-A) score greater than or equal to 10 at screening. Participants with anxiety disorder and/or mild major depressive disorder (with PHQ-A score ≤ 9) are permitted in the study if they are considered by the investigator to be stable and are taking no more than 1 medication for each disorder. Participant must have been on a stable dose within the 3 months before the start of the baseline phase.
  * Use of prohibited medication within 1 month before the start of the baseline phase and/or during the baseline phase.
  * Use of prohibited devices (such as stimulation devices) or procedures (such as acupuncture, biofeedback, relaxation techniques, or psychotherapy) with the goal of preventing migraines, within 3 months before the start of the baseline phase and/or during the baseline phase.
  * Participants receiving Cognitive Behavioral Therapy (CBT) are excluded unless they are on a stable, maintenance phase of a CBT program for migraine for at least 3 months before the start of the baseline phase. Participants undergoing CBT are considered on a stable, maintenance phase if they have undergone greater than or equal 6 weekly or biweekly sessions of CBT administered by adequately trained psychologists and who, for at least 3 months before the start of the baseline phase, only follow "booster" CBT sessions at a monthly, bimonthly or quarterly frequency. Note: Participants who have discontinued CBT within 3 months prior to the start of the baseline phase are eligible for the study provided that there is evidence of CBT failure/lack of efficacy prior to initial screening (per medical records or investigator's assessment).
  * Received botulinum toxin in the head and/or neck region within 4 months before the start of the baseline phase or during the baseline phase.
  * Received medication targeting the CGRP pathway within 4 months before the start of the baseline phase or during the baseline phase.
* Taken the following for any indication in any month during the 2 months before the start of the baseline phase, or during the baseline phase:

  * Ergotamines or triptans on greater than or equal 10 days per month.
  * Simple analgesics (nonsteroidal anti-inflammatory drugs [NSAIDs], acetaminophen) on greater than or equal 15 days per month.
  * Opioid or butalbital-containing analgesics on greater than or equal 4 days per month.
  * Currently receiving treatment in another investigational device or drug study, or less than 90 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
  * Participant has clinically significant vital signs, laboratory results, or ECG abnormality during screening that, in the opinion of the investigator, could pose a risk to participant safety or interfere with the study evaluation.
  * Hepatic disease by history or total bilirubin (TBL) greater than or equal 2.0 x upper limit of normal (ULN) or alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than or equal 3.0 x ULN, as assessed by the central laboratory at initial screening.
  * Female participant is pregnant or breastfeeding or planning to become pregnant or breastfeed during the study and for an additional 16 weeks after the last dose of investigational product. (Females of childbearing potential should only be included in the study after a confirmed menstrual period and a negative highly sensitive urine and serum pregnancy test.)
  * Female participants of childbearing potential unwilling to use an acceptable method of effective contraception during treatment and for an additional 16 weeks after the last dose of investigational product.
  * Participant has known sensitivity to any of the products or components to be administered during dosing.
  * Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant's legal representative and investigator's knowledge.
  * History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 457 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in MMDs | Baseline through week 12 of the double blind treatment phase
  To evaluate the effect of erenumab compared with placebo on the change in MMDs from baseline to week 9 through week 12 (month 3) of the double-blind treatment period (DBTP).

SECONDARY OUTCOMES:
Change in monthly headache days from baseline | Baseline through week 12 of the double blind treatment phase
  To evaluate the effect of erenumab compared with placebo on the change from baseline in monthly headache days to week 9 through week 12 (month 3) of the DBTP
Proportion of participants with at least 50% reduction in MMDs from baseline | Baseline through week 12 of the double blind treatment phase
  To evaluate the effect of erenumab compared with placebo on the proportion of participants with at least 50% reduction in MMDs from baseline to week 9 through week 12 (month 3) of the DBTP
Change in MMDs from baseline to the average of the first 3 months | Baseline through week 12 of the double blind treatment phase
  To evaluate the effect of erenumab compared with placebo on the change in MMDs from baseline to the average of the first 3 months (week 1 through week 12) of the DBTP
Change in monthly average severity of migraine attacks from baseline (measured with a visual analogue scale) | Baseline through week 12 of the double blind treatment phase
  To evaluate the effect of erenumab compared with placebo on the change from baseline in monthly average severity of migraine attacks to week 9 through week 12 (month 3) of the DBTP. This will be measured in a daily electronic diary (eDiary) with a visual analogue scale.
Change from baseline in migraine-related disability and productivity | Baseline through week 12 of the double blind treatment phase
  To evaluate the effect of erenumab compared with placebo on the change from baseline in migraine-related disability and productivity as measured by the modified PedMIDAS to week 9 through week 12 (month 3) of the DBTP.
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to week 80
  Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration will be recorded as TEAEs.
Change from baseline in C Terminal Telopeptide of Type 1 Collagen (CTX) Markers at assessment time points | Up to week 64
Change from baseline in Procollagen Type 1 N Propeptide (P1NP) Markers at assessment time points | Up to week 64
Number of Participants Expressing Anti-erenumab Antibodies | Up to week 80
Change in Growth and Development Rate as Assessed by Physical Measurements Based on Age-adjusted Z-scores for Height and Weight | Up to week 80
Number of Participants Experiencing Treatment-emergent Suicidal Ideation and Behavior as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to week 64
Group 1 Only: Number of Participants Experiencing Injection Site Pain as Assessed by Face Pain Scale-revised (FPS-R) | Day 1 and week 20
Group 2 Only: Number of Participants Experiencing Injection Site Pain as Assessed by FPS-R | Day 1 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (119):
- United States (38):
  - Paradigm Clinical Research Center Inc, San Diego, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Childrens National Health System, Washington D.C., District of Columbia
  - Northwest Florida Clinical Research Group Limited Liability Company, Gulf Breeze, Florida
  - Nicklaus Childrens Hospital, Miami, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - TrueBlue Clinical Research, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Rare Disease Research Center Pediatrics, Atlanta, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Chicago Headache Center and Research Institute, Chicago, Illinois
  - Josephson Wallack Munshower Neurology, Indianapolis, Indiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - New England Regional Headache Center Inc, Worcester, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute Inc, Minneapolis, Minnesota
  - Childrens Mercy Hospital and Clinics, Kansas City, Missouri
  - Mercy Research, St Louis, Missouri
  - Velocity Clinical Research, Inc, Grand Island, Nebraska
  - Dent Neurosciences Research Center, Amherst, New York
  - Modern Migraine MD, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Inc, Pittsburgh, Pennsylvania
  - Palmetto Gastroenterology Clinical Research, LLC, Summerville, South Carolina
  - Child Neurology Consultants of Austin, Austin, Texas
  - Helios Clinical Research Inc, Burleson, Texas
  - Stryde Consulting LLC, Frisco, Texas
  - Childrens Specialty Group, Norfolk, Virginia
  - Vaught Neurological Services, Crab Orchard, West Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - Algemeen Ziekenhuis Sint-Maarten, Mechelen
  - Docteur Simona Sava, Saint-Nicolas
- Canada (4):
  - Stollery Childrens Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital For Sick Children, Toronto, Ontario
- Colombia (7):
  - Fundacion Centro de Investigacion Clinica, Medellín, Antioquia
  - Servicios de Salud Ips Suramericana Sas - Ips Sura Industriales, Medellín, Antioquia
  - Institucion Prestadora de Servicios de Salud Sociedad Médica Rionegro SA Somer SA, Rionegro, Antioquia
  - Solano y Terront Servicios Medicos SAS - Unidad Integral de Endocrinologia Uniendo, Bogota, Cundinamarca
  - Cafam, Bogota, Cundinamarca
  - Fundacion Hospital Infantil Universitario De San Jose, Bogota, Cundinamarca
  - Fundacion cardiovascular de Colombia, Bucaramanga, Santander Department
- Terveystalo Pulssi, Turku, Finland
- Germany (5):
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Greifswald, Greifswald
  - Schmerzklinik Kiel, Kiel
  - Arzneimittelforschung Leipzig GmbH, Leipzig
- Hungary (6):
  - Dr Kenessey Albert Korhaz - Rendelointezet, Balassagyarmat
  - Dr Altmann Anna egyeni vallalkozo, Budapest
  - High Tech Medical Kft, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
- Italy (4):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda di Rilievo Nazionale e Alta Specializzazione Civico Di Cristina Benfratelli, Palermo
  - Fondazione Istituto Neurologico Nazionale C Mondino IRCCS, Pavia
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
- Japan (17):
  - Josai Kids Clinic, Nagoya, Aichi-ken
  - Medical Corporation Seikokai Takanoko Hospital, Matsuyama, Ehime
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Kitami Clinic, Sapporo, Hokkaido
  - Konan Medical Center, Kobe, Hyōgo
  - Umenotsuji Clinic, Kochi, Kochi
  - Kumamoto City Hospital, Kumamoto, Kumamoto
  - Tatsuoka Neurology Clinic, Kyoto, Kyoto
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto, Kyoto
  - Ishikawa Clinic, Kyoto, Kyoto
  - Sendai Headache and Neurology Clinic, Sendai, Miyagi
  - Tominaga Hospital, Osaka, Osaka
  - Saitama Neuropsychiatric Institute, Saitama-shi, Saitama
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Nagamitsu Clinic, Hofu-shi, Yamaguchi
  - Nagaseki Headache Clinic, Kai-shi, Yamanashi
- Poland (11):
  - Uniwersytecki Dzieciecy Szpital Kliniczny im Ludwika Zamenhofa w Bialymstoku, Bialystok
  - AthleticoMed, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Centrum Medyczne Luxmed Spzoo, Lublin
  - Centrum Medyczne Hope Clinic Sebastian Szklener, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Clinical Research Center Spzoo Medic-R Spolka Komandytowa, Poznan
  - Dr Sekowska Leczenie Bolu, Warsaw
  - Next Stage Spzoo, Warsaw
  - Migre Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
- Portugal (4):
  - Unidade Local de Saude de Coimbra, EPE - Hospital Pediatrico de Coimbra, Coimbra
  - Unidade Local de Saude de Sao Jose, EPE - Hospital Dona Estefania, Lisbon
  - Hospital da Luz, SA, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
- Puerto Rico Health and Wellness Institute, Dorado, Puerto Rico
- Russia (4):
  - FSBI Russian Children Clinical Hospital of the MoH RF, Moscow
  - LLC clinic Chaika, Moscow
  - LLC Sibneyromed, Novosibirsk
  - LLC Medical Technologies, Saint Petersburg
- Spain (5):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
- Switzerland (2):
  - Universitaets-Kinderspital beider Basel, Basel
  - Kopfwehzentrum Hirslanden, Zollikon
- United Kingdom (7):
  - Noahs Ark Childrens Hospital for Wales, Cardiff
  - Royal Hospital for Children, Glasgow
  - Alder Hey Childrens Hospital, Liverpool
  - Evelina Childrens Hospital, London
  - Great Ormond Street Hospital for Children, London
  - 4 Medical Clinical Solutions Manchester, Manchester
  - Oxford Childrens Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com